CLINICAL TRIAL: NCT01680003
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled Trial to Determine the Efficacy and Safety of HEPAR-P Capsule for the Treatment of Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Hepar-P Study to Evaluate the Safety and Efficacy of a Standardised Extract of Phyllanthus Niruri for the Treatment of Non-alcoholic Fatty Liver Disease
Acronym: Hepar-P
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nova Laboratories Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT11-03
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepar-P (Experimental): Hepar-P: Two capsules (250mg x 2), three times daily, orally
  Interventions: Drug: Hepar-P
- Placebo for Hepar-P (Placebo Comparator): Placebo: Two capsules, three times daily, orally
  Interventions: Drug: Placebo for Hepar-P

INTERVENTIONS:
Drug: Hepar-P
  Arms: Hepar-P
Drug: Placebo for Hepar-P
  Arms: Placebo for Hepar-P

SUMMARY:
This is a multi-center, double blind, parallel group placebo controlled randomised trial designed to determine the safety and efficacy of a Standardised Extract of Phyllanthus Niruri (EPN 797) HEPAR-P capsule for the treatment of Non-alcoholic Fatty Liver Disease for a treatment period of 48 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females age 18 years or older
* Written informed consent obtained from patient or parents/ guardian
* Elevated serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels but less than 2.5times the upper limit of the normal range
* Patients with liver biopsy confirmed possible or definite steatohepatitis within the past 12 months prior to enrolment into the trial
* Possible steatohepatitis with activity score ≥3 OR definite steatohepatitis with activity score ≥5
* A score of at least 1 for hepatocellular ballooning

Exclusion Criteria:

* Pregnant or nursing woman or women of childbearing potential except if post-menopausal, surgically sterile or using accepted method(s) of birth control or having negative pregnancy test
* Participation in any trial in which the patient received an investigational product within 30 days preceding the screening phase of this study
* Those persons directly involved in the conduct of the study
* Alcohol consumption of more than 20g per day for women or more than 30g per day for men for at least 3 consecutive months during the previous 5 years, as assessed with the use of the Lifetime Drinking History questionnaire and the interview version of the Alcohol Use and Disorders Identification Test (AUDIT)
* History of cirrhosis, hepatitis C or other liver diseases
* History of heart failure (New York Association Class II to IV)
* History of taking medications known to cause steatohepatitis
* Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in serum aspartate aminotransferase and alanine aminotransferase levels | 48 weeks

SECONDARY OUTCOMES:
Histologic findings including degree of steatosis, lobular inflammation, hepatocellular ballooning and fibrosis and overall disease activity score | 48 weeks

OTHER OUTCOMES:
Adverse events reporting, physical examinations and laboratory tests | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Radzi Abu Hassan, Dr, Principal Investigator — Sultanah Bahiyah Hospital, Alor Star; Tan Soek Siam, Dr, Principal Investigator — Selayang Hospital, Selangor; Tee Hoi Poh, Dr, Principal Investigator — Tengku Ampuau Afzan Hospital, Kuantan; Rosaida Mohd Said, Dr, Principal Investigator — Ampang Hospital, Selangor; Shashi Kumar Bhaskaran, Dr, Principal Investigator — Kuala Lumpur Hospital; Jayaram Menon, Dr, Principal Investigator — Queen Elizaberth Hospital, Sabah
Locations (5):
- Malaysia (5):
  - Sultamah Bahiyah Hospital, Alor Star, Kedah
  - Kuala Lumpur Hospital, Wilayah Persekutuan, Kuala Lumpur
  - Tengku Ampuan Afzan Hospital, Kuantan, Pahang
  - Queen Elizaberth Hospital, Kota Kinabalu, Sabah
  - Ampang Hospital, Kuala Selangor, Selangor